CLINICAL TRIAL: NCT04452123
Title: Endometrioma Treatment and Ovarian Function
Acronym: EnTOF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Jan Humplik, MD, Principal investigator, Charles University, Czech Republic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GPKENDO2001
Record Dates: First submitted 2020-06-12; First posted 2020-06-30 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Endometrioma
Keywords: Endometrioma; AMH
MeSH Terms: conditions — Endometriosis | interventions — Sutures

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Argon plasma (Experimental): Patients with endometrioma treated with laparoscopic argon plasma energy.
  Interventions: Procedure: Laparoscopic argon plasma treatment of endometrioma; Procedure: Laparoscopic stripping of endometrioma and suture/coagulation of the rest of ovary
- Stripping and suture/coagulation (Experimental): Patients with endometrioma treated with laparoscopic excision with suture or gentle coagulation of the rest of ovary.
  Interventions: Procedure: Laparoscopic argon plasma treatment of endometrioma; Procedure: Laparoscopic stripping of endometrioma and suture/coagulation of the rest of ovary

INTERVENTIONS:
Procedure: Laparoscopic argon plasma treatment of endometrioma — Laparoscopic Argon Plasma vaporising the endometriotic cyst lining only until haemosiderin pigment stained tissue is no longer visible
Procedure: Laparoscopic stripping of endometrioma and suture/coagulation of the rest of ovary — Laparoscopic dissecting of capsule of endometrioma and achieving hemostasis with suture of rest of the ovary or with gentle coagulation.

SUMMARY:
Ovarian endometriosis (endometrioma) can be a cause of subfertility. According to European Society of Human Reproduction and Embryology (ESHRE) guidelines, surgery for endometrioma is recommended when an endometrioma is more than 3 cm in diameter because this management is associated with better spontaneous conception rates. Nevertheless, surgery can also be potentially associated with a risk of destruction of functional ovarian tissue and reduction in ovarian reserve.

Anti-müllerian hormone (AMH) is a member of the Transforming Growth Factor beta family and is expressed by the small (<8 mm) pre-antral and early antral follicles. The AMH level reflects the size of the primordial follicle pool, and may be the best biochemical marker of ovarian function across an array of clinical situations Its level in serum is almost stable between 20 and 35 years of the woman´s life, unless using hormonal contraception and / or they suffer with Polycystic ovarian syndrome (PCOS). The level of AMH is also a useful indicator for the prediction chances of success of spontaneous or assisted conceptions. However, there paucity of data regarding changes in serum levels of AMH following surgery for endometrioma.

An alternative way for estimating ovarian reserve is quantifying ovarian mass with using standard 3D transvaginal ultrasound calculation (OVM) and assessment of antral follicular count.

The gold standard of endometrioma surgery is laparoscopic excision with suture or gentle coagulation of the rest of ovary or by the use of laparoscopic treatment with argon plasma energy.

ELIGIBILITY:
Inclusion Criteria:

* women with endometrioma 3cm and more in diameter

Exclusion Criteria:

* using hormonal contraception or other hormonal treatment last 6 months
* suffer with polycystic ovarian syndrome

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
AMH | 3 days,3-5 week postop., 3 months postop., 1 year (optional)
  Changing of anti-müllerian hormon assay postop. in µg/L
Antral follicle count (AFC) | 3 months, 1 year
  Ultrasound count of Antral follicles after the surgery, counted 3-5. day of menstrual cycle
Both ovarian volume | 3 months, 1 year
  Ultrasound volume of both ovaries in cm^3, measured 3-5. day of menstrual cycle

CONTACTS AND LOCATIONS:
Overall Officials: Jan Humplik, MD, Principal Investigator — Charles university in Pilsen
Locations (1):
- Departement of gynecology and obstetrics, University hospital in Pilsen, Pilsen, Czechia

IPD SHARING:
Plan to Share IPD: No